CLINICAL TRIAL: NCT00100256
Title: Open Label Study of Single Dose Rhenium Re 188 P2045 in Patients With Lung Cancer Who Have Received or Refused to Receive Prior Chemotherapy
Brief Title: Rhenium Re 188 P2045 in Patients With Lung Cancer Who Have Received or Refused to Receive Prior Chemotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andarix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91168; 306509
Record Dates: First submitted 2004-12-27; First posted 2004-12-28 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Neoplasm Recurrence, Local
Keywords: Advanced or recurrent stage IIIb or IV non small cell lung cancer; Disseminated or recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Neoplasm Recurrence, Local; Small Cell Lung Carcinoma | interventions — Rhenium

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Rhenium (Re 188 P2045, BAY86-5284)

INTERVENTIONS:
Drug: Rhenium (Re 188 P2045, BAY86-5284) — Infusion once only

SUMMARY:
The purpose of this study is to determine the maximum dose that is safely tolerated of the experimental drug Rhenium Re 188 P2045. This will be done by first treating patients at relatively low doses of Rhenium Re 188 P2045, observing them closely to assure that there are no bad side effects, then increasing the dose when we are confident that it is safe to do so.

DETAILED DESCRIPTION:
We want to learn more about the side effect profile of both Technetium Tc 99m P2045 and Rhenium Re 188 P2045 and will do that by observing you closely after you receive the drug and by conducting multiple tests, as well as by asking you how you feel. We want to also learn if there is any benefit, in terms of lung cancer tumor reduction, as a result of treatment with Rhenium Re 188 P2045. This study has previously been posted by Berlex, Inc. Andarix Pharmaceuticals is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically documented Non-Small-Cell Lung Cancer (NSCLC) or Small-Cell Lung Cancer (SCLC) and has advanced or recurrent IIIb or IV NSCLC (adenocarcinoma, squamous cell carcinoma, large cell, mixed or not otherwise specified) or disseminated or recurrent SCLC or any lung cancer which has local recurrence.
* Has documentation of progressive disease following prior chemotherapy or who refused to receive standard chemotherapy.
* Has measurable tumor (at least 1 cm unidimensionally) in a previously non-irradiated area or, if in previously irradiated area, a substantial increase in size of tumor, based on CT scan within 8 weeks prior to enrollment; tumor in previously irradiated area only if it has increased by 50% or more from previous minimal diameter AND it is more than 8 weeks from the radiation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-01; Primary Completion 2009-06-20 (Actual); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of Rhenium 188 P2045 | Over the first month post dose administration
  Toxicity as determined by the analysis protocol
Safety of Technetium Tc 99m P2045 and Rhenium Re 188 P2045 | Up to one year post study completion
  Examination of clinical chemistry indicators as outlined in the protocol
Progression free survival in treated patients | Up to one year post study completion
  Analyze tumor and disease progression after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Andarix Study Director, Study Director — Andarix Pharmaceuticals
Locations (2):
- United States (2):
  - Iowa City, Iowa
  - Baltimore, Maryland